CLINICAL TRIAL: NCT06236802
Title: ProVIDE II Bridging Study for the ProVee System for BPH
Brief Title: ProVIDE II Bridging Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ProVerum Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP 003
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: BPH With Symptomatic Lower Urinary Tract Symptoms
Keywords: BPH / LUTS
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- ProVee treatment (Experimental): ProVee Expander is placed in prostatic urethra to relieve obstruction due to BPH.
  Interventions: Device: ProVee device

INTERVENTIONS:
Device: ProVee device — ProVee Expander is placed in prostatic urethra to relieve obstruction due to BPH.
  Other Names: ProVee Expander; ProVee

SUMMARY:
The purpose of the ProVIDE II Bridging Study is to evaluate the performance of the Generation II delivery system when deploying the ProVee expander in subjects with symptomatic urinary obstruction secondary to BPH.

DETAILED DESCRIPTION:
This is a prospective, multi-center, open-label, non-randomized bridging study to evaluate the performance of the Generation II delivery system when deploying the ProVee expander in subjects with symptomatic urinary obstruction secondary to benign prostatic hyperplasia (BPH).

ELIGIBILITY:
Inclusion Criteria:

1. Males > 45 years of age
2. IPSS of ≥ 13, IPSS V/S > 1 at baseline assessment
3. Prostate volume of ≥ 30 cc and ≤ 80 cc
4. Prostatic urethral L2 lengths ≥ 3.75 cm by TRUS
5. Failed, intolerant, or subject choice to not take a medication regimen for the treatment of LUTS.

Exclusion Criteria:

1. Void volume <125 ml; Qmax > 12 ml/s; PVR > 250 ml
2. Obstructive median lobe defined by EITHER >10mm protrusion on sagittal mid-prostate plane as measured by TRUS OR an obstructive median lobe seen on cystoscopy e.g., 'ball valve''
3. High bladder neck, with the absence of lateral lobe encroachment indicating a high likelihood of primary bladder neck obstruction
4. Anatomy that would prevent the apices of the ProVee from engaging with the lateral lobes e.g., high degree of bladder neck angulation such that the anterior bladder neck is not visible
5. Acute urinary retention
6. Known immunosuppression
7. History of or suspected prostate or bladder cancer
8. Baseline PSA > 10 ng/mL or confirmed or suspected prostate cancer (Subjects with a PSA level above 2.5 ng/mL, or age specific, or local reference ranges should have prostate cancer excluded to the Investigator's satisfaction, including a SOC biopsy if indicated).
9. Recent urinary tract stones OR widespread calcifications on the prostatic urethral wall, within 3 months of index procedure
10. A history of prostatitis within the last two years
11. Active or history of epididymitis within the past 3 months
12. Neurogenic bladder and/or sphincter abnormalities due to Parkinson's disease, multiple sclerosis, cerebral vascular accident, diabetes
13. History of urinary retention within 12 months of baseline assessment
14. Requiring self-catheterization to void
15. An active urinary tract infection (UTI) at time of index procedure
16. Gross haematuria, within 3 months of index procedure.
17. Subjects with known allergy to nickel or titanium
18. Life expectancy estimated to be less than 60 months
19. Taking androgens, unless eugonadal state for at least 3 months or greater with a stable dosage for at least 2 months as documented by the Investigator
20. Use of 5-alpha-reductase inhibitors (e.g., dutasteride, finasteride) within 6 months of baseline assessment
21. Use of Phenylephrine / Pseudoephedrine within 24 hours of baseline assessment
22. Use of alpha-blockers (e.g., Terazosin, Doxazosin, Alfuzosin, Tamsulosin) within 2 weeks of baseline assessment
23. Use of estrogen or drug-producing androgen suppression (e.g. gonadotropin-releasing hormonal analogues) within 1 year of baseline assessment
24. Use of antihistamines, anticonvulsants, and antispasmodics within 1 week of baseline assessment unless there is documented evidence that the patient was on the same drug dose for at least 6 months with a stable voiding pattern (the drug dose should not be altered or discontinued for entrance into or throughout the study)
25. Use of anticholinergics or cholinergic medication within 2 weeks of baseline assessment
26. Use of beta-blockers where the dose is not stable. (Stable dose is defined as having the same medication and dose in the last 6 months)
27. Use of Phosphodiesterase-5 Enzyme Inhibitors in doses for BPH within 2 weeks of baseline assessment.
28. Current treatment with anticoagulants (e.g., coumadin or enoxaparin) or antiplatelet medications other than aspirin (e.g., clopidogrel, or alternative and ASA). Patient unable to stop taking anticoagulants and/or antiplatelets within 3 days prior to the procedure or coumadin at least 5 days prior to the procedure. Low dose aspirin ≤100mg/day not prohibited
29. Future fertility concerns
30. Previous prostate surgery, balloon dilatation, stent implantation, laser prostatectomy, hyperthermia, or any other invasive treatment to the prostate; including penile implants
31. Previous pelvic irradiation or radical pelvic surgery
32. Previous rectal surgery (other than haemorrhoidectomy) or known history of rectal disease
33. Urethral strictures, bladder neck contracture, or other potentially confounding bladder pathology
34. Urethral pathologies that may prevent insertion of Delivery System
35. Uncontrolled diabetes mellitus including Hgb AIC >8%
36. Overactive bladder (OAB) requiring treatment by OAB medication
37. Urinary incontinence
38. Patients taking tri-cyclic antidepressants.
39. Compromised renal function (i.e., serum creatinine >1.8 mg/dl or upper tract disease)
40. Hepatic disorder, bleeding disorders or metabolic impairment that might confound the results of the study or have a risk to subject per investigator's opinion
41. Any major comorbidities or presence of unstable conditions, e.g., uncontrolled HTN, NYHA Class III or IV, cardiac arrhythmias that are not controlled by medication/medical device, myocardial infarction within the past 6 months, COPD with FEV1 <50, renal illness that might prevent study completion or would confound study results
42. Vulnerable populations such as incarcerated or institutionalized adults, inmates, patients with physical, psychological (such as developmentally delayed adults), or medical impairment that might, in the judgment of the Investigator, prevent study completion or comprehension, or may confound study results (including patient questionnaires)
43. History or current medical condition that would result in an unacceptable patient risk if that subject were to be included in the study
44. Any subject that is currently enrolled in another ongoing investigational study.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 40 (Actual)
Dates: Start 2024-03-06 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Events | (time frame: procedure to 3 months)
  Rate of device or procedure related serious adverse events through 3-months.
Need for urinary catheterization | (time frame: >7 days post procedure to 3-months)
  The rate of extended post-operative urinary catheterization (> 7 days from treatment) for inability to void among patients treated with the ProVee System for BPH.
Technical Success | Procedure
  The percentage of subjects where the expander is deployed in the location intended by the user. This endpoint will be met if the Observed Technical Success is >95%.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (7):
  - Florida Urology Partners, LLP, Tampa, Florida
  - Avant Concierge Urology, Winter Garden, Florida
  - Comprehensive Urologic Care, Lake Barrington, Illinois
  - Sheldon Freeman MD LTD, Las Vegas, Nevada
  - Midtown Urology Assoc. PA, Austin, Texas
  - Urology Austin, Austin, Texas
  - Houston Methodist Research Institute, Houston, Texas
- St James Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data (IPD) available to other researchers

REFERENCES:
- See also: ProVerum Website — https://www.proverummedical.com/